CLINICAL TRIAL: NCT04011007
Title: Comparison of Vitrectomy Without Internal Limiting Membrane Peeling Versus Inverted ILM Flap Technique for Macular Hole Retinal Detachment in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31241
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Macular Holes; Retina Detachment
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitrectomy without ILM peeling (Active Comparator): vitrectomy without ILM peeling
  Interventions: Procedure: vitrectomy with or without inverted ILM flap technique
- vitrectomy with inverted ILM flap technique (Active Comparator): vitrectomy with inverted ILM flap technique
  Interventions: Procedure: vitrectomy with or without inverted ILM flap technique

INTERVENTIONS:
Procedure: vitrectomy with or without inverted ILM flap technique — vitrectomy without ILM peeling versus vitrectomy with inverted ILM flap technique in cases of macular hole retinal detachment in high myopic eyes.

SUMMARY:
The aim of this study was to determine whether inverted ILM peeling technique could contribute to high reattachment and closure rates after vitrectomy in patients with myopic macular hole retinal detachment (MHRD) in comparison to no ILM peeling.

This retrospective study will include 40 patients presenting by myopic macular hole retinal detachment. Exclusion criteria will include history of trauma, choroidal neovascularization, and the presence of a peripheral retinal break or proliferative vitreoretinopathy before the initial surgery.

Subjects will be divided into 2 groups; Group 1 will include 20 patients that were treated by vitrectomy without ILM peeling and postoperative gas or silicone oil tamponade with or without cataract surgery.

Group 2 will include 20 patients that were treated by vitrectomy with ILMflap technique and postoperative gas or silicone oil tamponade with or without cataract surgery.

ELIGIBILITY:
Inclusion Criteria: macular hole retinal detachment in high myopic eyes.

-

Exclusion Criteria:

* eyes with previous vitreoretinal surgery, trauma, diabetic retinopathy, retinal vein occlusion, uveitis, and other retinal diseases were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
visual acuity at one year | 12 months

SECONDARY OUTCOMES:
rate of retinal attachment and macular hole closure. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt